CLINICAL TRIAL: NCT00196664
Title: Assessment of the Efficacy of Paroxetine in the Prevention of Depressive Syndrome in Patients With Chronic Hepatitis C Treated by PEG-Interferon Alfa Plus Ribavirin. Multicentric, Double-Blinded, Randomized Study. ANRS HC18 Paropeg
Brief Title: Efficacy of Paroxetine in the Prevention of Depressive Syndrome in Patients With Chronic Hepatitis C Treated by PEG-Interferon Alfa Plus Ribavirin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-004102-24; ANRS HC18 PAROPEG
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Paroxetine; Depression
MeSH Terms: conditions — Hepatitis C, Chronic; Depression | interventions — Paroxetine

INTERVENTIONS:
Drug: Paroxetine

SUMMARY:
Depression is a common side effect of interferon in the treatment of chronic hepatitis C. The aim of this study is to assess the efficacy and safety of paroxetine, an antidepressant agent, in the prevention of depression induced by PEG-interferon given for the treatment of chronic hepatitis C.

DETAILED DESCRIPTION:
The aim of this study is to assess the efficacy and safety of paroxetine, an antidepressant agent, in the prevention of depression induced by PEG-interferon given for the treatment of chronic hepatitis C. This is a comparative study including two groups of patients randomly allocated : one with paroxetine and the other with the placebo. The rate of depression will be compared between the 2 groups

ELIGIBILITY:
Inclusion Criteria:

- Chronic hepatitis C which should be treated by PEG-interferon alfa and ribavirin with no contra-indication to anti-viral treatment

Exclusion Criteria:

* Allergy to paroxetine
* Current antidepressant treatment
* Depression diagnosed by the MINI International Neuropsychiatric Interview (MINI, DSM IV)
* History of bipolar syndrome
* History of psychotic syndrome
* Treatment by triptan, carbamazepine, millepertuis, methadone, oral anticoagulation
* Renal insufficiency
* HIV infection
* Breath feeding
* Contra-indication to PEG-interferon and or ribavirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2005-10; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Incidence of depression based on MINI International Neuropsychiatric Interview (MINI, DSM IV)from D0 to W74

SECONDARY OUTCOMES:
Evolution of depression score (MADRS and BDI scales) to W74,Quality of life (HQL questionnaire), Fatigue, Compliance to PEG-interferon and ribavirin, Virological response at W74 ,Safety

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre Bronowicki, MD, PhD, Principal Investigator — Service d'Hépato-gastroenterologie, CHU de Nancy, Vandoeuvre France; Faiez Zannad, MD, Study Chair — C.I.C Nancy France
Locations (1):
- Service d'Hépato-gastroentérologie CHU de Nancy, Vandœuvre-lès-Nancy, France